CLINICAL TRIAL: NCT05570903
Title: A Prospective Observational Cohort Study of Awake Prone Position Ventilation Strategy in Patients With Acute Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yuan-Qiang Lu, Professor, First Affiliated Hospital of Zhejiang University
Other Study IDs: luyuanqiang
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Awake prone position Group: Patients in awake prone position will be included.
- Non awake prone position Group: Patients in non awake prone position will be included.

SUMMARY:
Awake prone positioning has been used widely for patients with COVID-19.Many research results are not uniform on the key issue of whether the prognosis of patients can be improved，and most of the subjects were patients with SARS-CoV-2 infected who are not intubated.The investigators will conduct a prospective observational study on patients with acute respiratory failure induced by various causes to determine whether awake prone position can reduce the need to upgrade to invasive mechanical ventilation and improve the prognosis of patients compared with standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.Older than 17 years, admitted to the ICU;2.Patients with acute respiratory failure meet the following conditions：①Under the condition of breathing air at rest, PaO2 of subjects is lower than 60mmHg and/or PaCO2 is higher than 50mmHg; ②Under the support of COT and HFNC, PaO2/FiO2 of the subject is less than 250; ③ Under the support of NIV ;

Exclusion Criteria:

* 1.Refusing to cooperate with active treatment; 2.Immediate need for intubation as determined by the treating team.3Patients with hemodynamic instability and moderate to high dose of vasopressors (norepinephrine dose ≥ 0.15 mcg/kg/min)；4.Contraindication to PP (e.g. vomiting, abdominal wound, unstable pelvic/spinal lesions, pregnancy >20/40 gestation, severe brain injury)；

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute and critical patients transferred from primary hospitals or admitted to emergency departments
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2024-10-09 (Estimated); Study Completion 2025-09-09 (Estimated)

PRIMARY OUTCOMES:
Endotracheal intubation rate | 28 days
  Percentage of patients in each group whose respiratory support means are upgraded to endotracheal intubation
Mortality | 28 days
  Death

SECONDARY OUTCOMES:
Total hours of prone position at day | 28 days
  Total hours of prone position at day
Total number of prone sessions at day | 28 days
  Total number of prone sessions at day
Total days of prone positioning therapy | 28 days
  Total days of prone positioning therapy
Non-invasive ventilation days | 28 days
  Number of days not receiving non-invasive mechanical ventilation
Change in the ROX-index 1-hour after first prone session | 1 hour
  The change in the Ratio of SpO2/FiO2 to respiratory rate (ROX-index)
Total length of stay in ICU and hospital | 28 days
  Total length of stay in ICU and hospital